CLINICAL TRIAL: NCT01724320
Title: A Phase I, First-in-man Study of OTX008 Given Subcutaneously as a Single Agent to Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oncoethix GmbH, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTX008_101
Record Dates: First submitted 2012-11-02; First posted 2012-11-09 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Solid Tumors
Keywords: solid tumors; first-in-man; phase I; cancer; galectin
MeSH Terms: conditions — Neoplasms | interventions — compound 0118

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OTX008 (Experimental): Single-arm study of OTX008 given subcutaneously, daily without interruption to patients with advanced solid tumors. Starting dose: 65 mg/day.
  Interventions: Drug: OTX008

INTERVENTIONS:
Drug: OTX008 — OTX008 given daily without interruption, subcutaneously. Starting dose: 65 mg/day

SUMMARY:
The purpose of this study is to determine the recommended dose (RD) for further phase II studies, of the Galectin-1 inhibitor OTX008 given subcutaneously in patients with advanced solid tumors

DETAILED DESCRIPTION:
Overexpression of galectin-1 protein is well documented in different types of cancers, with associated bad prognostic and enhanced metastases spreading.

In-vitro/in-vivo preclinical studies showed that OTX008 inhibits galectin-1 expression. In different cancer models in animals, OTX008 reduced tumor growing and metastases spreading and it was observed a blood vessels architecture normalization.

Thus, OTX008 appears to be an innovating approach to treat cancers and this clinical phase I study aims to evaluate OTX008 therapy in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to beginning protocol specific screening procedures. Patients registered in this trial must be treated and followed at the participating centers. Patients should receive the study treatment within 7 days after registration
* Histologically proven malignant solid tumor
* Patients having failed all standard therapies, or for whom standard therapies are deemed ineffective or contra-indicated.
* Patients aged > 18 years.
* ECOG performance status (PS) of 0 to 1
* Off previous systemic therapy (except LH-RH agonist therapy started > 2 months prior to study entry that could be continued) , radiation therapy, or surgery for at least 30 days prior to first study treatment administration (45 days for bicalutamide).
* Recovery from the toxic effects of prior treatment to NCIC-CTC grade < 1, except alopecia
* Adequate bone marrow function including: Neutrophils >= 1.5 x 10E9 /L; platelets >= 100 x 10E9 /L, Hb > 8g/dL without transfusion.
* Creatinine clearance >= 60 mL/min (Cockroft & Gault formula, or MDRD formula for patients aged > 65 years).
* Adequate LFTs: Total bilirubin < 1 x the institutional upper normal limits (UNL); ALAT/ASAT >= 3 x UNL (or >= 5 x UNL in case of liver metastases).
* Serum albumin > 28g/L.
* Availability of the last tumor imaging within 6 months prior to baseline tumor imaging
* Availability of archived pathology specimen (paraffin-embedded block) from the tumor

Exclusion Criteria:

* History of prior malignancy other than those previously treated with a curative intent more than 5 years ago and without relapse (any tumor) or basal cell skin cancer, in situ cervical cancer, superficial bladder cancer, or high grade intestinal polyps treated adequately, regardless of the disease-free interval.
* Pregnant or lactating women or women of childbearing potential not using adequate contraception. Male patients not using adequate contraception.
* Tumor sites that necessitate immediate intervention (supportive care, surgery or radiation therapy) such as symptomatic brain or leptomeningeal tumor, spinal cord compression, other compressive tumor masses, painful bone metastasis, bone fracture, etc…
* Other serious illness or medical conditions, which, in the investigator's opinion could jeopardize patient's safety or hamper understanding of the study by the patient, patient's compliance to study treatment, or interpretation of study results. These conditions include (but are not restricted to):

  1. Congestive heart failure or angina pectoris not medically controlled. Previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or arrhythmias.
  2. Existence of significant neurologic or psychiatric disorders impairing the ability to obtain consent.
  3. Active infection.
* Concurrent treatment with other experimental therapies or participation in another clinical trial within 30 days prior to first study treatment administration.
* Concurrent treatment with any other anticancer therapy (except LH-RH agonist therapy initiated > 2 months prior to study entry).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | up to 3 weeks of OTX008 treatment
  Dose Limiting Toxicity (DLT) will be assessed during the first 21 days (3 weeks)of OTX008 treatment in each patient to determine Recommended Dose (RD)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Days 1, 2 and 22 of OTX008 treatment
  OTX008 plasma concentration will be assessed at days 1, 2 and 22 of OTX008 treatment to determine PK profile of OTX008. Following parameters will be used: Trough (Cmin) and peak (Cmax) of OTX008 concentrations, Tmax, t1/2, steady state, total clearance, AUC (Area Under Curve)
Pharmacodynamics (PD) | Days 1 and 22 of OTX008 treatment
  Following parameter will be measured: plasma levels of galectin-1

CONTACTS AND LOCATIONS:
Locations (3):
- Institut Jules Bordet, Brussels, Belgium
- France (2):
  - Hopital Beaujon - AP-HP, Clichy
  - Institut Claudius Regaud, Toulouse